CLINICAL TRIAL: NCT05010343
Title: Functional Image-Guided Carbon Ion Irradiation With Simultaneous Integrated Boost for Prostate Cancer: a Phase II Randomized Controlled Clinical Trial
Brief Title: Functional Image-Guided Carbon Ion Irradiation With Simultaneous Integrated Boost for Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Proton and Heavy Ion Center (Other)
Responsible Party: Principal Investigator, Ping Li, Principal Investigator, Shanghai Proton and Heavy Ion Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPHIC-TR-PCa2020-01
Record Dates: First submitted 2021-03-14; First posted 2021-08-18 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Localized Prostate Cancer
Keywords: carbon ion irradiation; Simultaneous Integrated Boost; PSMA PET/CT; mpMRI

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- carbon ion irradation group (Active Comparator): All patients will receive carbon ion irradiation with 65.6 GyE in 16 fractions to the prostate with or without seminal vesicle
  Interventions: Radiation: carbon ion irradation
- Carbon Ion Irradiation With SIB group (Active Comparator): All patients will receive carbon ion irradiation with 65.6 GyE in 16 fractions to the prostate with or without seminal vesicle, and with simultaneous integrated boost (SIB) to the gross tumor in the PSMA PET/CT and mpMRI
  Interventions: Radiation: Carbon Ion Irradiation With SIB

INTERVENTIONS:
Radiation: carbon ion irradation — All patients will receive carbon ion irradiation with 65.6 GyE in 16 fractions to the prostate with or without seminal vesicle
  Arms: carbon ion irradation group
Radiation: Carbon Ion Irradiation With SIB — All patients will receive carbon ion irradiation with 65.6 GyE in 16 fractions to the prostate with or without seminal vesicle, and with simultaneous integrated boost (SIB) to the gross tumor in the PSMA PET/CT and mpMRI
  Arms: Carbon Ion Irradiation With SIB group

SUMMARY:
This is a phase II randomized controlled clinical trial to assess the toxicities and clinical efficacy of prostate specific membrane antigen (PSMA) positron emission tomography / computed tomography (PET/CT) and multi- parameter Magnetic Resonance Imaging (MRI) guided simultaneous integrated boost for prostate cancer.

DETAILED DESCRIPTION:
Local recurrences of prostate cancer following radiotherapy often originate from the primary tumor site. Therefore,focal boost to the primary gross tumor has been proposed to increase biochemical disease-free survival (bDFS) without increasing toxicity.

The higher relative biological effectiveness (RBE) and greater cytocidal effect on the intrinsic radiation resistant cancer cells offer carbon ion radiotherapy (CIRT) advantages over conventional radiotherapy. In this study, carbon ion were used to treat localized prostate cancer and simultaneous integrated boost to the gross tumor in the prostate specific membrane antigen (PSMA) PET/CT and multi- parameter MRI.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed adenocarcinoma of prostate
* Stage cT1-3N0M0 localized prostate cancer
* performed PSMA PET/CT and mpMRI before treatment
* No lymph nodes or distant metastasis
* Age ≥ 45 and < 85 years of age
* Karnofsky Performance Score ≥70
* No previous pelvic radiation therapy (RT)
* No previous prostatectomy
* No previous invasive cancer (within 5 years before the prostate cancer diagnosis)
* Ability to understand character and individual consequences of the clinical trial
* Willing to sign the written informed consent; Informed consent must be signed before the enrollment in the trial

Exclusion Criteria:

* No pathologically confirmed adenocarcinoma of the prostate
* Pelvic lymph node metastasis (N1)
* Distant metastasis (M1)
* Previous pelvic radiotherapy
* Previous prostatectomy

Ages: 45 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2020-10-15 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Acute toxicities | Within 3 months of the start of CIRT
  Treatment related acute toxicity assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 4.03

SECONDARY OUTCOMES:
Late toxicities | 3 months after the completion of CIRT
  Treatment related late toxicity assessed by Radiation Therapy Oncology Group (RTOG) scale
Biochemical failure free survival | From the complation of CIRT,a median of 5 years
  The prostate specific antigen less than nadir plus 2ng/ml (Phoenix definition)
Overall survival | From the diagnosis of prostate cancer,a median of 5 years
  The time from diagnosis to death from any cause
Progression free survival | From the complation of CIRT,a median of 5 years
  The time from complation of CIRT to tumor progression or death

OTHER OUTCOMES:
The quality of life-International Prostate Symptom Score (IPSS) | From the complation of CIRT, a median of 5 years
  IPSS would be used to assess the severity of lower urinary tract symptoms, based on the answers to seven questions regarding urinary symptoms (incomplete emptying, frequency, intermittency, urgency, weak stream, straining, and nocturia).
  Total IPSS score: 1-7: Mild; 8-19: Moderate; 20-35: Severe
The quality of life-Expanded Prostate Cancer Index Composite (EPIC) | From the complation of CIRT, a median of 5 years
  EPIC would be used to evaluate the urinary, bowel, and sexual symptoms. The EPIC is a patient reported outcomes instrument designed to evaluate bowel, urinary, sexual and hormonal domains both during and after irradiation of the pelvis.For each domain, responses are provided on a 5-point Likert scale, and multi-item scale scores are transformed linearly to a scale of 0 to 100, where higher scores correspond to better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Proton and Heavy Ion Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hu W, Li P, Hong Z, Guo X, Pei Y, Zhang Z, Zhang Q. Functional imaging-guided carbon ion irradiation with simultaneous integrated boost for localized prostate cancer: study protocol for a phase II randomized controlled clinical trial. Trials. 2022 Nov 8;23(1):934. doi: 10.1186/s13063-022-06798-5. PMID 36348363